CLINICAL TRIAL: NCT06917560
Title: The Role of Serological Autoantibody Profiles in the Early Diagnosis and Prognosis of Renal Carcinoma: A Multicenter, Retrospective Clinical Study
Brief Title: Serological Autoantibodies in Early Kidney Cancer Diagnosis and Prognosis: A Multicenter Study
Status: Active, not recruiting | Type: Observational
Sponsor: First Affiliated Hospital of Fujian Medical University (Other)
Collaborators: China-Japan Friendship Hospital (Other); The First Affiliated Hospital of Xiamen University (Other)
Responsible Party: Sponsor
Other Study IDs: MRCTA,ECFAH OfFMUI2024]697
Record Dates: First submitted 2025-04-01; First posted 2025-04-08 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: Renal Carcinoma; Serology; Autoantibody
Keywords: Renal Carcinoma; Autoantibody; serology
MeSH Terms: conditions — Carcinoma, Renal Cell

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This project aims to construct a multicenter retrospective study by retrospectively collecting clinical, serological, and pathological data from patients. A comprehensive data management system will be established to facilitate the integration and analysis of multicenter data, alongside antibody profiling characteristics. A predictive model based on serological autoantibody profiles will be developed and validated using both internal and external cohorts. This model will predict clinical prognostic factors in renal carcinoma and identify patient populations likely to respond to immunotherapy. By enabling personalized treatment decisions and minimizing unnecessary treatment risks, the model aims to improve patient quality of life and overall prognosis.

ELIGIBILITY:
Inclusion Criteria:

* Pathological diagnosis of ccRCC;
* Availability of complete clinical, pathological, and follow-up data;
* Sufficient preoperative serum available for collection;
* Well-preserved pathological slides for subsequent immunohistochemical (chip) analysis;
* At least one post-treatment follow-up/efficacy evaluation.

Exclusion Criteria:

* Therapeutic contraindication cohort: Individuals presenting with severe comorbidities rendering them medically ineligible for therapeutic interventions;
* Oncological multiplicity: Subjects with either (a) antecedent therapeutic regimens targeting non-index malignancies or (b) concurrent diagnosis of untreated active malignancies;
* Biospecimen integrity violation: Cases demonstrating serum hemolysis or compromised specimen integrity;
* Data insufficiency cohort: Patients exhibiting incomplete clinical/pathological records or insufficient longitudinal follow-up data for comprehensive analysis.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients with histologically confirmed renal cell carcinoma
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2025-04-01 (Actual); Primary Completion 2027-08-01 (Estimated); Study Completion 2027-08-01 (Estimated)

PRIMARY OUTCOMES:
serum autoantibodies | Prior to any treatment or surgery, 5 mL of venous blood was collected from each individual and allowed to stand at room temperature (RT) for 1 hour to facilitate coagulation.
  After incubating the serum on the HuProt array, autoantibody signals were detected, standardized, and quantified. For the selection of candidate proteins, three criteria must be met when comparing ccRCC with healthy controls: (1) a p-value ≤ 0.05 obtained from the t-test; (2) a fold change (FC) ≥ 1.2; (3) a positivity rate ≥ 10% (ccRCC positive reactivity is defined as values greater than the average of the healthy control group plus 2× SD. The positivity rate is calculated as the ratio of ccRCC positive responses to the total number of responses).

CONTACTS AND LOCATIONS:
Locations (1):
- first hospital affiliated of Fujian medical university, Fuzhou, Fujian, China

IPD SHARING:
Plan to Share IPD: Undecided